CLINICAL TRIAL: NCT01534923
Title: Doctor-Patient Communication About Colorectal Cancer Screening
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Albert Einstein College of Medicine (Other); HHC, Gun HIll and Tremont (Unknown); NYC RING, Director (Unknown); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Other Study IDs: 12-017
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Colorectal Cancer Screening
Keywords: Doctor-Patient Communication; questionnaire; survey; 12-017
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Pts having colorectal cancer screening: The target sample of this study will be approximately 200 primary care physician-patient consultations who discuss CRC screening during the course of a clinical visit. Physician and patient participants will come from primary care practices associated with the New York City Research and Improvement Networking Group (NYC RING).
  Interventions: Behavioral: surveys

INTERVENTIONS:
Behavioral: surveys — The intervention will be the audio-recording of the physician-patient consultation, patient and doctor surveys. These audio recordings will be coded. It will also include follow-up phone calls with patients.

SUMMARY:
The purpose of this study is to learn more about doctor-patient communication about colon cancer screening. This study will also look to see if there are differences in those who get colon cancer screening based on the discussion the doctor had with the patient.

ELIGIBILITY:
Inclusion Criteria:

Physicians

* Attending physicians or third year residents specializing in internal medicine or family medicine, as per the medical director from the clinic.
* Clinic is based at a NYC RING-affiliated practice.
* English speaking; Due to limited resources, we cannot have each audio recorded consultation translated therefore, the consultation needs to be in English.

Patients

* Ages 50-75 years old, per the United States Preventive Services Task Force recommendations for screening. This will be determined by a pre-screening of medical records by the RSA.
* Due for colorectal cancer screening at the time of the visit, ascertained through patient self-report (e.g., no colonoscopy within the past 10 years, no flexible sigmoidoscopy or barium enema within the past five years, and no FOBT within the past year).
* Coming for either an annual physical exam or chronic care follow up visit, per patient self-report.
* Planning to consult with the physician in English, per patient self-report. Due to limited resources, we cannot have each audio recorded consultation translated therefore, the consultation needs to be in English.

Exclusion Criteria:

* History of colorectal cancer, per patient self-report or per EMR..
* History of polyps being removed, per patient self-report.
* Colonoscopy scheduled in EMR at time of screening.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Five health centers of the NYC RING will participate in this project. All are located in underserved urban communities within the Bronx.
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2012-02-07 (Actual); Primary Completion 2019-12-26 (Actual); Study Completion 2019-12-26 (Actual)

PRIMARY OUTCOMES:
describe doctor-patient communication about CRC screening | 2 years
  screening adherence through self report. Screening adherence will be assessed by contacting the patients and asking them if they received the CRC screening test their doctor ordered at the audio recorded visit.

SECONDARY OUTCOMES:
quality of doctor-patient communication about CRC screening and low-income patients' screening outcomes. | 2 years
examine the association between the quality of doctor-patient communication about CRC screening and low-income patients' screening outcomes | 2 years
  intent to be screened (immediately after the consultation) using the item from Geller et al.25 and 2) self-efficacy for screening (immediately after consultation) in case there are few events of actual screening.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Ostroff, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Albert Einstein College of Medicine, The Bronx, New York
  - Hhc, Gun Hill and Tremont, The Bronx, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/